CLINICAL TRIAL: NCT00799669
Title: Cancer Risk Reduction Through Combined Treatment for Tobacco and Alcohol Use
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000626365; MDA-2005-0791; CDR0000626365 (Other: NCI Clinical Trials); U54CA096300 (NIH); U54CA096297 (NIH); NCI-2012-02110 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer; Tobacco Use Disorder
Keywords: hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; tobacco use disorder
MeSH Terms: conditions — Head and Neck Neoplasms; Tobacco Use Disorder; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Counseling; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MAPS+: MAPS+ (Motivation and Problem-Solving Plus):
  Counseling using specific treatment approach that focuses on combined smoking cessation and the reduction of at-risk alcohol use.
  Interventions: Behavioral: smoking cessation intervention; Other: counseling intervention; Other: preventive intervention; Other: questionnaire administration
- MAPS: MAPS (Motivation and Problem-Solving):
  Counseling treatment approach with a focus on smoking cessation.
  Interventions: Behavioral: smoking cessation intervention; Other: questionnaire administration

INTERVENTIONS:
Behavioral: smoking cessation intervention — Standard quit-smoking counseling to help decrease their risk of cancer.
Other: counseling intervention — Counseling focusing on decreasing risk of getting cancer by decreasing smoking and alcohol use.
  Groups: MAPS+
Other: preventive intervention
  Groups: MAPS+
Other: questionnaire administration
  Other Names: survey

SUMMARY:
RATIONALE: A counseling program that motivates patients to stop smoking and drinking may reduce the risk of oral cancer. It is not yet known whether motivational stop smoking counseling or motivational stop-smoking and stop drinking counseling is more effective in helping patients stop smoking and drinking.

PURPOSE: This randomized clinical trial is studying how well treatment to stop smoking and drinking works in preventing oral cancer in smokers in Puerto Rico.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effects of a motivational and problem-solving smoking cessation (MAPS) and a motivational and problem solving approach on at-risk alcohol use and smoking cessation (MAPS+) among Puerto Rican at-risk drinkers/smokers who call the Puerto Rico Quitline (PRQ).
* To assess effects of MAPS and MAPS+ on treatment mechanisms and the role of those mechanisms in mediating these effects on at-risk drinking and smoking cessation.
* To evaluate the cost-effectiveness of MAPS and MAPS+ in the reduction of at-risk drinking and smoking cessation.

OUTLINE: Minimization randomization is applied using the following variables: age, gender, cigarettes/day, number of drinks/day, and depression (score on the Center of Epidemiologic Studies Depression Scale). Patients are randomized to 1 of 2 intervention arms.

* Arm I (MAPS): Patients receive culturally sensitive self-help materials tailored for alcohol and tobacco users and 7 telephone counseling calls. The MAPS approach includes motivational interviewing and cognitive behavioral/problem-solving that focus on smoking cessation.
* Arm II (MAPS+): Patients receive culturally sensitive self-help materials tailored for alcohol and tobacco users and 7 telephone counseling calls. The MAPS+ approach includes motivational interviewing and cognitive behavioral/problems solving that focus on smoking cessation and the reduction of at-risk alcohol use.

In both arms, patients receive counseling calls over 15-30 minutes the week before quit date (QD), on QD, 3-5 days after QD, 7-10 days after QD, 15-30 days after QD, 45-60 days after QD, and on day 90 after QD. Patients complete questionnaires for alcohol- and smoking-related measures, self efficacy, stress/negative affects/depression, social support, and physical activity at baseline and weeks 12, 26 and 52 after QD.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current daily smoker
* Called the Puerto Rico Quitline
* Motivated to quit smoking in the next 30 days
* Exhibits at least one of the following criteria for at-risk drinking:

  * An average of ≥ 2 alcoholic beverages/day for men or ≥ 1 drink/day for women in the past 30 days
  * Two or more occasions of consuming ≥ 5 alcoholic beverages/day for men or ≥ 4 drinks/day for women in the past 30 days
  * Driving after consuming ≥ 3 drinks in the past 30 days
* Score of ≤ 15 on the Alcohol Use Disorders Identification Test

PATIENT CHARACTERISTICS:

* Not pregnant
* Residing in Puerto Rico
* Not currently incarcerated or in jail
* No other household member enrolled in this study
* Viable telephone number and home address
* Willing to provide the names, addresses, and phone numbers of up to 3 collaterals

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Smokers Residing in Puerto Rico
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2007-12-05 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Participant At-risk drinking status | 52 weeks
Smoking cessation | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PhD, MS, BA, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org
- See also: National Cancer Institute (NCI) Central Website for Cancer Research — http://www.cancer.gov/about-cancer/treatment/clinical-trials/search?